CLINICAL TRIAL: NCT00050193
Title: Determining the Pathogenesis of Systemic Pediatric-Onset Mastocytosis
Brief Title: Cause and Natural Course of Pediatric-Onset Mastocytosis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030041; 03-I-0041
Record Dates: First submitted 2002-11-25; First posted 2002-11-26 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-03-10

CONDITIONS: Mastocytosis
Keywords: Children; Mast Cells; Urticaria Pigmentosa; Bone Marrow; Severe; Mastocytosis; Pediatric Mastocytosis
MeSH Terms: conditions — Mastocytosis; Urticaria Pigmentosa; Lymphoma, Follicular

SUMMARY:
This study will evaluate children with mastocytosis, a disease of excessive mast cells in tissues such as skin and bone marrow, to identify the cause of the disease and describe its course. Mast cells can release chemicals that cause itching, blisters, flushing, bone pain, and abdominal pain. Usually, mastocytosis in children involves the skin only and is of limited duration. This study, however, will focus on children with more severe disease that more closely resembles adult-onset mastocytosis.

Patients up to 21 years of age with childhood-onset mastocytosis may be eligible for this study. Candidates must have one or more of the following abnormalities, which indicate severe disease: enlarged liver or spleen; diffuse skin involvement; history of gastrointestinal bleeding or peptic ulcer; bone marrow biopsy with abnormal mast cells either in number or shape; elevated blood levels of the enzyme tryptase; or abnormal hemoglobin, white blood cells, platelets, or clotting factors.

Participants will have a medical history and physical examination; various blood tests, including studies to identify genetic changes that are important in the growth, development, and functioning of human mast cells; and bone marrow aspiration and biopsy. For the bone marrow procedure, the skin over the hipbone and the outer surface of the bone itself are numbed with an injection of local anesthesia. Then, a special needle is inserted into the hipbone and about 2 tablespoons of bone marrow are drawn into a syringe. Another needle is then inserted through the first needle to collect a small piece of the bone marrow. Pain will be managed according to the individual patient s needs. Additional procedures, such as a gastroenterology consultation, colonoscopy to examine the colon, or computerized axial tomography (CT) or ultrasound of the abdomen to assess the liver and spleen, may be done if medically indicated. Standard medical treatment, including antihistamines for itching or steroids for abdominal cramping or diarrhea, will be recommended as appropriate.

Patients biologic parents may also be enrolled to provide a blood sample for genetic analysis and a bone marrow aspirate and biopsy for clinical and research purposes.

Patients will return to NIH once a year for follow-up evaluations until their disease is stable or until the 5-year study ends.

...

DETAILED DESCRIPTION:
Mastocytosis in infants and children is an unusual disease characterized by an excess of mast cells in tissues. In pediatric onset mastocytosis, disease is usually localized to the skin and disease is considered to be of limited duration. However, a subset of children appear to develop a clinical picture resembling that observed in adults who have adult-onset disease. This study will focus on children with more severe mastocytosis in an attempt to define its pathogenesis, focusing on mutations and polymorphisms in genes regulating mast cell proliferation and survival to determine if they might contribute to this disease pattern. If severe pediatric-onset disease does not fit within the existing classification, new criteria of diagnosis must be proposed for the pediatric age group.

This study will examine children and young adults age birth to 21 years with pediatric-onset disease previously enrolled on NIAID mastocytosis protocols, or as a result of physician referral, which have disease more consistent with adult-onset disease or parameters associated with increased morbidity. The evaluation may include serum tryptase, blood count, bone marrow biopsy and aspirate, morphology and mutational analysis. Subjects may be asked to return in 12-24 months for assessment. If relevant mutation effecting mast cell growth and function are identified, such mutations will be sought in the biologic parents as appropriate, but only when such mutations are believed to be germ line (not somatic) mutations. This study will aid in the understanding of the characteristics of severe mastocytosis in the pediatric age group.

ELIGIBILITY:
* INCLUSION CRITERIA:

Children with tissue-diagnosed pediatric-onset mastocytosis formerly enrolled in protocols 90-I-0120, and 93-I-0136 or per physician referral with more severe disease as indicated by one of the following parameters:

* Hepatomegaly or splenomegaly;
* Diffuse cutaneous mastocytosis;
* History of gastrointestinal bleeding or peptic ulcer disease;
* Bone marrow biopsy with abnormal numbers or shaped mast cells or abnormal flow cytometry;
* Serum tryptase greater than 20ng/ml;
* Hematologic abnormalities such as an increase WBC, thrombocytosis, and/or an increase in PT and/or PTT.

INCLUSION CRITERIA-SUBJECT:

* Age birth to 21.0 years of age at the time of entry into the protocol
* Diagnosis of mastocytosis by skin examination or histologic evidence in a skin or bone marrow biopsy
* Subject has a primary medical care provider outside the NIH
* Subject or parent or guardian is able to give informed consent

INCLUSION CRITERIA-RELATIVE:

* A biological relative with or without the diagnosis of mastocytosis by skin examination or histologic evidence in a skin or bone marrow biopsy
* Subject has a primary medical care provider outside the NIH

EXCLUSION CRITERIA SUBJECT:

* Age greater than or equal to 21.0 years
* No primary care physician
* Has AIDS or is HIV Positive

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2002-11-22; Study Completion 2014-03-10

CONTACTS AND LOCATIONS:
Overall Officials: Melody C Carter, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kettelhut BV, Metcalfe DD. Pediatric mastocytosis. Ann Allergy. 1994 Sep;73(3):197-202; quiz 202-7. PMID 8092552
- [Background] Kirshenbaum AS, Goff JP, Kessler SW, Mican JM, Zsebo KM, Metcalfe DD. Effect of IL-3 and stem cell factor on the appearance of human basophils and mast cells from CD34+ pluripotent progenitor cells. J Immunol. 1992 Feb 1;148(3):772-7. PMID 1370517
- [Background] Dvorak AM, Seder RA, Paul WE, Morgan ES, Galli SJ. Effects of interleukin-3 with or without the c-kit ligand, stem cell factor, on the survival and cytoplasmic granule formation of mouse basophils and mast cells in vitro. Am J Pathol. 1994 Jan;144(1):160-70. PMID 7507298